CLINICAL TRIAL: NCT01537393
Title: Effect of Corneal Preservation Time on Long-Term Graft Success
Brief Title: Cornea Preservation Time Study
Acronym: CPTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Eye Institute (NEI) (NIH); Jaeb Center for Health Research (Other)
Responsible Party: Principal Investigator, Jonathan Lass, MD, Charles I Thomas Professor, Dept. of Ophthalmology & Visual Sciences,, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPTS; 1U10EY020798-01A1 (NIH); 1U10EY020797-01A1 (NIH)
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Cornea Preservation Time; Endothelial Keratoplasty; Transplant Success; Endothelial Cell Density
Keywords: cornea; transplant; preservation; endothelial keratoplasty
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0-7d Preservation Time Group (Other): Subjects in this arm will receive cornea tissue transplant with cornea tissue preserved for 0 to 7 days prior to transplant.
  Interventions: Biological: Cornea tissue transplant
- 8-14d Preservation Time Group (Other): Subjects in this arm will receive cornea tissue transplant with cornea tissue preserved for 8 to 14 days prior to transplant.
  Interventions: Biological: Cornea tissue transplant

INTERVENTIONS:
Biological: Cornea tissue transplant — Cornea tissue preserved 0 to 7 days
  Arms: 0-7d Preservation Time Group
Biological: Cornea tissue transplant — Cornea tissue preserved 8 to 14 days.
  Arms: 8-14d Preservation Time Group

SUMMARY:
The purpose of this study is to determine if the 3-year graft failure rate following endothelial keratoplasty performed with donor corneas with a preservation time of 8 to 14 days is non-inferior to the failure rate when donor corneas with a preservation time of 7 or fewer days are used.

DETAILED DESCRIPTION:
When the donor cornea is removed from the person who died, it is prepared for transplantation by an eye bank. The donor cornea is placed into a liquid that helps preserve the cornea until it is transplanted. The Food and Drug Administration (FDA) has approved storage of the cornea in this liquid for up to 14 days before the transplant. The purpose of this study is to see if the length of time the donor cornea is kept in the preservation liquid before the transplant affects the likelihood of the transplant being successful. We will follow participants for 3 years after transplant to see if there are any differences in transplant success or in the number of transplanted endothelial cells (the layer of cells that line the undersurface of the cornea) on the corneas that were preserved for 7 days or less compared to those preserved between 8 and 14 days. We have no reason to believe that there is any greater risk for transplant failure with either preservation time group.

ELIGIBILITY:
Study Participant Eligibility Criteria

* Study Participant Inclusion Criteria

  1. Age range 30-<91 years with minimum life expectancy of at least 3 years.
  2. Willingness to return for follow-up study visits at 1 day, 1 week, 1 month, 6 months, 1 year, 2 years and 3 years.
  3. Fluent in English or Spanish.
* Study Participant Exclusion Criteria 1) Decisionally and/or cognitively impaired

Study Eye Eligibility Criteria

* Study Eye Inclusion Criteria

  1. Endothelial keratoplasty (EK) is scheduled between 10 and 60 days after enrollment

     * The 10-day requirement relates to the need to be able to randomly assign the eye to either intervention group.
     * The 60-day requirement relates to the need to have current eligibility and enrollment data at the time of surgery. If surgery is postponed to >60 days after the initial enrollment visit, a new Baseline Visit and eligibility assessment will have to be performed.
  2. Presence of a condition related to endothelial dysfunction which will be treated by EK.
* Eligible indications for EK include:

  * Presence of Fuchs endothelial corneal dystrophy (FECD) meeting at least one of the following:

    * Phakic FECD
    * Phakic FECD with cataract

      * Triple procedure including EK for FECD, cataract extraction and posterior chamber intraocular lens implantation (IOL) is allowed
    * Aphakic FECD
    * Pseudophakic FECD with posterior capsule supported, suture-fixated, or sulcus-supported posterior chamber IOL
  * Aphakic or pseudophakic corneal edema with posterior capsule supported, suture-fixated, or sulcus-supported posterior chamber IOL without FECD
* Study Eye Exclusion Criteria

  1. Prior EK
  2. Indication for surgery that is not suitable for EK (e.g, keratoconus, stromal dystrophies and scars)
  3. Presence of a condition that has a very high probability for failure (e.g., failed EK or Penetrating Keratoplasty (PKP), heavily vascularized cornea, uncontrolled uveitis)
  4. Other primary endothelial dysfunction conditions including posterior polymorphous corneal dystrophy and congenital hereditary corneal dystrophy
  5. Anterior chamber IOL in study eye prior to or anticipated during EK
  6. Planned intraocular lens exchange of an anterior chamber IOL with a posterior chamber IOL in study eye at time of study EK
  7. Pre-operative central sub-epithelial or stromal scarring that the investigator believes is visually significant and could impact post-operative stromal clarity assessment
  8. Stromal vascularization that is visually significant (by investigator's judgment)
  9. Presence of anterior synechiae (iris to cornea)
  10. Peripheral anterior synechiae (iris to angle) in the angle greater than a total of three clock hours
  11. Hypotony (Intraocular pressure <10 mm Hg)
  12. Uncontrolled (defined as intraocular pressure > 25mm Hg) glaucoma with or without prior filtering surgery or shunt or mini-shunt placement.

      * A shunt or mini-shunt is any device implanted to lower intraocular pressure through an external route (e.g Ahmed) or internal route (e.g. Glaukos) that is present in the anterior chamber angle or extends into the anterior chamber.
  13. Controlled glaucoma with prior shunt or mini-shunt placement for glaucoma

      * Note: FECD or pseudophakic/aphakic corneal edema with posterior chamber IOL that also have undergone filtering surgery (without shunt or mini-shunt) in which glaucoma is currently considered under control will be eligible
  14. Fellow eye visual acuity < 20/200 that is not correctable with EK

Eligibility Criteria for Second Study Eye

1. Study participant has already enrolled one eye
2. The second eye meets all study eye inclusion and exclusion criteria (2.2.2 and 2.2.3)
3. EK surgery in second eye is not planned within 6 weeks of EK on first study eye

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1174 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lass, MD, Study Chair — Case Western Reserve University; Allison Ayala, MS, Principal Investigator — Jaeb Center for Health Research
Locations (40):
- United States (40):
  - Keck Medical Center, Beverly Hills, California
  - Jules Stein Eye Institute, Los Angeles, California
  - Eye Care of San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Center for Sight, Sarasota, Florida
  - Woolfson Eye Institute, Atlanta, Georgia
  - Eye Consultants of Atlanta, Atlanta, Georgia
  - University of Illinois Eye and Eye, Chicago, Illinois
  - NorthShore University Health System, Glenview, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky Ophthalmology, Lexington, Kentucky
  - Mid-Atlantic Cornea Consultants, Baltimore, Maryland
  - Johns Hopkins/Wilmer Eye Institute, Baltimore, Maryland
  - Eye Consultants of Maryland, Owings Mills, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - University of Michigan/Kellogg Eye Center, Ann Arbor, Michigan
  - Verdier Eye Center, Grand Rapids, Michigan
  - Michigan Cornea Consultants, Southfield, Michigan
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mercy Medical Research Institute, Springfield, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Cornea Consultants of Albany, Slingerlands, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - University Hospitals Case Medical Center Eye Institute, Cleveland, Ohio
  - Ohio State Medical Center, Columbus, Ohio
  - Northeast Ohio Eye Surgeons, Kent, Ohio
  - Medical Eye Center, Medford, Oregon
  - Devers Eye Institute, Portland, Oregon
  - Ophthalmic Partners of PA, Bala-Cynwyd, Pennsylvania
  - Central Pennsylvania Eye Institute, Hershey, Pennsylvania
  - Sadeer Hannush, MD, Langhorne, Pennsylvania
  - Corneal Associates, PC, Wills Eye Institute, Philadelphia, Pennsylvania
  - Cornea Associates of Texas, Dallas, Texas
  - Focal Point Vision, San Antonio, Texas
  - University of Utah, Moran Eye Center, Salt Lake City, Utah
  - Eye Associates Northwest, Seattle, Washington
  - Dean Medical Center, Madison, Wisconsin

REFERENCES:
- [Result] Rosenwasser GO, Szczotka-Flynn LB, Ayala AR, Liang W, Aldave AJ, Dunn SP, McCall T, Navarro LC, Pramanik S, Ross KW, Stulting RD, Terry MA, Tu EY, Verdier DD, Kollman C, Gal RL, Beck RW, Lass JH; Cornea Preservation Time Study Group. Effect of Cornea Preservation Time on Success of Descemet Stripping Automated Endothelial Keratoplasty: A Randomized Clinical Trial. JAMA Ophthalmol. 2017 Dec 1;135(12):1401-1409. doi: 10.1001/jamaophthalmol.2017.4989. PMID 29127431
- [Result] Lass JH, Benetz BA, Verdier DD, Szczotka-Flynn LB, Ayala AR, Liang W, Aldave AJ, Dunn SP, McCall T, Mian SI, Navarro LC, Patel SV, Pramanik S, Rosenwasser GO, Ross KW, Terry MA, Kollman C, Gal RL, Beck RW; Cornea Preservation Time Study Group. Corneal Endothelial Cell Loss 3 Years After Successful Descemet Stripping Automated Endothelial Keratoplasty in the Cornea Preservation Time Study: A Randomized Clinical Trial. JAMA Ophthalmol. 2017 Dec 1;135(12):1394-1400. doi: 10.1001/jamaophthalmol.2017.4970. PMID 29127432
- [Derived] Lass JH, Bailey RJ, Szczotka-Flynn LB, Benetz BA, Soper M, Titus MS, Kollman C, Beck RW; Cornea Preservation Time Study Group. Comparison of Graft Outcomes Reusing Original Intermediate-Term Cold Storage Solution for Entire Corneal Donor Storage Period With Exchanged Fresh Storage Solution After Donor Preparation in the Cornea Preservation Time Study. Cornea. 2022 Dec 1;41(12):1539-1544. doi: 10.1097/ICO.0000000000003108. Epub 2022 Sep 9. PMID 36036663
- [Derived] Lass JH, Szczotka-Flynn LB, Ayala AR, Benetz BA, Gal RL, Aldave AJ, Corrigan MM, Dunn SP, McCall TL, Pramanik S, Rosenwasser GO, Ross KW, Terry MA, Verdier DD; Writing Committee for the Cornea Preservation Time Study Group. Cornea preservation time study: methods and potential impact on the cornea donor pool in the United States. Cornea. 2015 Jun;34(6):601-8. doi: 10.1097/ICO.0000000000000417. PMID 25850706
- See also: Public website — http://cpts.jaeb.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was at eye level. When both eyes of a participant were included, the eye undergoing surgery 1st was assigned randomly to a PT group and the 2nd eye to the other group. 2 eyes had their assigned donor corneas inadvertently switched, and resulted in 1 of these participants receiving both study eyes from 8-14d group.
Units Other Than Participants: eyes
Groups:
- 0-7d Preservation Time (PT) Group: Subjects in this arm will receive cornea tissue preserved for up to 7 days prior to transplant.
  Cornea tissue transplant: Cornea tissue preserved either 7 or less days or 8 to 14 days.
- 8-14d Preservation Time (PT) Group: Subjects in this arm will receive cornea tissue preserved for 8 to 14 days prior to transplant.
  Cornea tissue transplant: Cornea tissue preserved either 7 or less days or 8 to 14 days.
Period: Overall Study
Arm/Group | 0-7d Preservation Time (PT) Group | 8-14d Preservation Time (PT) Group
Started (1046 eyes from 1151 participants randomized) | 707; 707 eyes | 698; 699 eyes
Completed (Study eyes with 3-year visit completed) | 553; 553 eyes | 507; 508 eyes
Not Completed | 154; 154 eyes | 191; 191 eyes
Not completed — Exclude prior to study | 32 | 44
Not completed — Death | 20 | 32
Not completed — Withdrawal by Subject | 18 | 17
Not completed — Lost to Follow-up | 53 | 48
Not completed — Failure - Regrafted | 28 | 43
Not completed — Failure - Not regrafted | 2 | 6
Not completed — Censored (severe event unrelated to PT) | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analyses conducted at eye level. 1330 study eyes of 1090 participants underwent descemet stripping automated endothelial keratoplasty. 480 eyes completed bilateral surgery (240 participants), 1 participant had both eyes received cornea in 8-14 days group. 435 and 414 participants underwent unilateral surgery in 0-7 and 8-14 days groups.
Units Other Than Participants: eyes
Groups:
- Preservation Time Group 1: Subjects in this arm will receive cornea tissue preserved for up to 7 days prior to transplant.
  Cornea tissue transplant: Cornea tissue preserved either 7 or less days or 8 to 14 days.
- Preservation Time Group 2: Subjects in this arm will receive cornea tissue preserved for 8 to 14 days prior to transplant.
  Cornea tissue transplant: Cornea tissue preserved either 7 or less days or 8 to 14 days.
- Total: Total of all reporting groups
Arm/Group | Preservation Time Group 1 | Preservation Time Group 2 | Total
Number analyzed (Participants) | 675 | 654 | 1090
Number analyzed (eyes) | 675 | 655 | 1330
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [64 to 76] | 70 [64 to 77] | 70 [64 to 76]
Sex: Female, Male [Count of Units; unit: eyes]
  Female | 409 | 392 | 801
  Male | 266 | 263 | 529
Race/Ethnicity, Customized [Count of Units; unit: eyes]
  White | 613 | 594 | 1207
  African American | 26 | 21 | 47
  Hispanic or Latino | 19 | 25 | 44
  Asian | 7 | 5 | 12
  American India or Alaskan Native | 1 | 2 | 3
  More than 1 race | 6 | 3 | 9
  Unknown or not reported | 3 | 5 | 8
History of Diabetes [Count of Units; unit: eyes] | 116 | 126 | 242
Current cigarette smoker [Count of Units; unit: eyes] | 45 | 45 | 90
Received any immunizations or vaccinations in last 3 mo [Count of Units; unit: eyes] | 92 | 81 | 173
Prior glaucoma surgery [Count of Units; unit: eyes] | 18 | 13 | 31
Glaucoma medication currently being used [Count of Units; unit: eyes] | 45 | 54 | 99
Diagnosis [Count of Units; unit: eyes]
  Pseudophakic corneal edema without FECD | 44 | 29 | 73
  Aphakic corneal edema without FECD | 0 | 2 | 2
  Fuchs endothelial corneal dystrophy (FECD) | 631 | 624 | 1255
Corneal Dystrophy other than FECD (Fuchs endothelial corneal dystrophy)) [Count of Units; unit: eyes] — During the slit lamp exam performed using the investigator's usual routine, the presence of other corneal dystrophies was recorded; EBMD=epithelial basement membrane dystrophy
  eyes
    No | 630 | 623 | 1253
    Keratoconus | 1 | 0 | 1
    EBMD (epithelial basement membrane dystrophy) | 38 | 29 | 67
    Other | 6 | 3 | 9
Stromal corneal vessels present (but not visually significant) [Count of Units; unit: eyes] | 4 | 1 | 5
Central subepithelial/stromal scarring present (not affect postoperative stromal clarity assessment) [Count of Units; unit: eyes] | 37 | 48 | 85
Peripheral anterior synechiae present (nongonioscopic) [Count of Units; unit: eyes] | 4 | 2 | 6
Preoperative lens status [Count of Units; unit: eyes] — During the slit lamp exam performed using the investigator's usual routine, the state of the crystalline lens was described as phakic (present), aphakic (removed), or pseudophakic (removed with posterior chamber intraocular lens inserted)
  eyes
    Phakic | 341 | 351 | 692
    Aphakic | 0 | 2 | 2
    Pseudophakic posterior chamber intraocular lens | 334 | 302 | 636
Postoperative lens status [Count of Units; unit: eyes]
  Phakic | 4 | 6 | 10
  Pseudophakic posterior chamber intraocular lens | 671 | 649 | 1320
Intraocular pressure (IOP) [Median (Inter-Quartile Range); unit: mm Hg] | 15 [12 to 17] | 15 [12 to 17] | 15 [12 to 17]

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With Corneal Graft Failure Within 3 Years of Surgery
Description: Graft failure, defined as the occurrence of one of the following within 3 years of surgery:
  * Regrafting of the study eye for any reason
  * Cornea which remains cloudy without clearing, according to the following:
    1. cloudy cornea on the first postoperative day which does not clear within 8 weeks OR
    2. cloudy cornea which was initially clear postoperatively but becomes and remains cloudy for 3 months without clearing.
Time Frame: Study eye will be assessed for this outcome for 3 years following surgery
Population: Analyzed number of eyes in each group (Overall 1090 unique participants)
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Preservation Time Group 1 | Preservation Time Group 2
Number analyzed (Participants) | 675 | 654
Number analyzed (Eyes) | 675 | 655
Eyes | 30 | 49
Statistical Analysis 1: Comparison: Preservation Time Group 1 vs Preservation Time Group 2; Test type: Non-Inferiority — The two treatment groups will be declared equivalent if the one-sided 95% confidence interval for the difference in proportions excludes the pre-defined non-inferiority limit of 4%; Risk Difference (RD) = 3.2, 95% CI 1-sided [upper limit 5.4]; The bootstrap re-sampling technique were used to account for potentially correlated data from donors who donated both corneas in this study and potentially correlated data from 2 study eyes of the same study participant. The technique will sample with replacement from the observed dataset. Confidence intervals will be calculated using the bias-corrected and accelerated method. The number of bootstraps will be 100,000
Statistical Analysis 2: Comparison: Preservation Time Group 1 vs Preservation Time Group 2; Test type: Other — Confounding and treatment interactions were assessed in Cox proportional hazards regression models; p = 0.02, Regression, Cox; Unadjusted Hazard Ratio; Hazard Ratio (HR) = 1.71, 95% CI 2-sided [1.09 to 2.71]

2. Primary Outcome: Endothelial Cell Density (ECD)
Description: Endothelial cell density at 3 years from surgery, conditional on graft survival at 3 years from surgery.
Time Frame: 3 years from surgery
Population: Eyes with graft success and a gradable image at 3 year (945 eyes of 769 unique participants)
Measure: Mean (Standard Deviation); unit: Cells per square millimeter
Units Other Than Participants: eyes
Arm/Group | Preservation Time Group 1 | Preservation Time Group 2
Number analyzed (Participants) | 485 | 459
Number analyzed (eyes) | 485 | 460
Cells per square millimeter | 1722 (626) | 1642 (631)
Statistical Analysis 1: Comparison: Preservation Time Group 1 vs Preservation Time Group 2; Test type: Other — The primary analysis to assess the effect of PT on 3 year ECD was conducted with a mixed linear model adjusting for baseline ECD, corneal diagnosis, and potential confounders, including storage solution, preparation by eye bank vs surgeon, and accounting for correlated data from participants with 2 study eyes or 2 corneas from the same donor; p = 0.03, Mixed Models Analysis; Adjusted for baseline ECD, diagnosis, storage solution, preparation by eye bank/surgeon, participants with 2 study eyes/ 2 corneas from the same donor; Mean Difference (Final Values) = 73, 95% CI 2-sided [8 to 138]

ADVERSE EVENTS:
Time Frame: Through study completion, up to 5 years
Description: Adverse event was collected at eye level
Groups:
- 0-7d Preservation Time Group: Subjects in this arm will receive cornea tissue preserved for up to 7 days prior to transplant.
  Cornea tissue transplant: Cornea tissue preserved either 7 or less days or 8 to 14 days.
- 8-14d Preservation Time Group: Subjects in this arm will receive cornea tissue preserved for 8 to 14 days prior to transplant.
  Cornea tissue transplant: Cornea tissue preserved either 7 or less days or 8 to 14 days.
Arm/Group | 0-7d Preservation Time Group | 8-14d Preservation Time Group
All-Cause Mortality (participants affected / at risk) | 20/675 | 32/654
Serious Adverse Events (participants affected / at risk) | 1/675 | 2/654
Other Adverse Events (participants affected / at risk) | 0/675 | 0/654
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0-7d Preservation Time Group (N=675) | 8-14d Preservation Time Group (N=654)
Endophthalmitis (Eye disorders) | 1 | 0 — One case of bacterial endophthalmitis occurred in the 0-7d PT group 4 days after surgery
Microbial keratitis (Eye disorders) | 0 | 2 — Microbial keratitis (bacterial, fungal, parasitic) within 3 months of endothelial keratoplasty (EK) 2 cases of fungal keratitis occurred in the 8-14d PT group 13 and 43 days after surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT01537393/Prot_SAP_000.pdf